CLINICAL TRIAL: NCT02520882
Title: Safety and Diagnostic Performance of 68Gallium-labeled NOTA-Aca-BBN(7-14) PET/CT in Patients With Primary Gliomas
Brief Title: 68Ga-NOTA-Aca-BBN(7-14) PET/CT in Patients With Primary Gliomas
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM11; ZIAEB000073 (NIH)
Record Dates: First submitted 2015-08-02; First posted 2015-08-13 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2015-03

CONDITIONS: Glioma
Keywords: PET/CT; Bombesin; gastrin-releasing peptide receptor; 68Gallium labeling
MeSH Terms: conditions — Glioma | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-Aca-BBN(7-14) PET/CT (Experimental): The patients were injected with 111-148 MBq of 68Ga-NOTA-Aca-BBN(7-14) in one dose intravenously and underwent PET/CT scan 30 min later.
  Interventions: Drug: 68Ga-NOTA-Aca-BBN; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-NOTA-Aca-BBN — 68Ga-NOTA-Aca-BBN(7-14) were injected into the patients before the PET/CT scans
  Other Names: 68Ga-NOTA-Aca-BBN(7-14)
Device: PET/CT

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-Aca-BBN(7-14) in glioma patients. A single dose of 111-148 Mega-Becquerel (MBq) 68Ga-NOTA-Aca-BBN(7-14) will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
Non-invasive imaging evaluation of GRPR expression would be of great help in drug development, patient stratification and therapeutic response monitoring. Various GRPR targeting imaging probes have been develop to meet the purpose. Bombesin (BBN) is an amphibian homolog of mammalian gastrin-releasing peptide (GRP). BBN(7-14), with the amino acid sequence of Gln-Trp-Ala-Val-Gly-His-Leu-Met-NH2, has been extensively used for the development of molecular probes for the imaging of gastrin-releasing peptide receptor (GRPR), after being labeled with various radionuclides. Multiple preclinical studies have demonstrated receptor-specific accumulation of the tracers in GRPR positive tumors. For interests in clinical translation of 68Ga-NOTA-Aca-BBN(7-14), an open-label dynamic whole-body PET/ CT study was designed to investigate the safety and diagnostic performance of 68Ga-NOTA-Aca-BBN(7-14) in patients with glioma.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Clinically based and magnetic resonance imaging (MRI)-based suspected newly diagnosed primary glioma.
* The tumor will be surgically removed and histological diagnosis will be available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential；
* Known severe allergy or hypersensitivity to IV radiographic contrast；
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-Aca-BBN(7-14) in primary glioma | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in primary glioma will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, Dr., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No